CLINICAL TRIAL: NCT06635681
Title: Efficacy of Venetoclax Combined with Intensive Chemotherapy in Different Subgroups of Acute Myeloid Leukemia : a Multi-center, Single-arm Clinical Trial
Brief Title: Efficacy of Venetoclax Combined with Intensive Chemotherapy in Different Subgroups of AML
Acronym: DAV-AML-2024
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024074
Record Dates: First submitted 2024-09-27; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: AML (Acute Myelogenous Leukemia)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Antineoplastic Combined Chemotherapy Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- venetoclax combined with intensive chemotherapy (Experimental): Induction therapy: daunorubicin, cytarabine, combined with venetoclax for 1 course.
  Consolidation therapy: cytarabine combined with venetoclax for 3 courses.
  Maintenance therapy: azacitidine combined with venetoclax for 6 courses.
  Interventions: Drug: combined chemotherapy

INTERVENTIONS:
Drug: combined chemotherapy — Induction therapy(1 cycle):
  Daunorubicin 60mg/m2/d d1-3 Cytarabine 100mg/m2/d d1-7 Venetoclax 100mg d-2, 200mg d-1, 400mg d1-7 If the first course of treatment did not result in CR, patients with therapeutic target could be treated with targeted drugs, and the patients without targets would be treated with HAV regimen: Cytarabine 100mg/m2/d, d1-5, Homoharringtonine 2mg/m2 d1-5, Venetoclax 100mg d-2, 200mg d-1, 400mg d1-7.
  Consolidation therapy(3 cycles):
  Cytarabine 2g/m2 q12h d1-3 Venetoclax 400mg d1-7 For patients with CBF and CEBPA dual mutations, the dose of cytarabine is 3g/m2.
  Maintenance treatment(6 cycles):
  Azacitidine 75mg/m2/d d1-5 Venetoclax 400mg d1-7
  Allogeneic hematopoietic stem cell transplantation is recommended for high-risk groups and intermediate-risk with positive measurable residual disease.

SUMMARY:
Acute myeloid leukemia (AML) is a common hematological malignancy. Intensive chemotherapy is the main treatment in fit patients.

Retrospective studies have shown that Venetoclax is highly effective in elder AML patients with IDH2 and NPM1 mutations while in those with TP53 and FLT3 mutations, the combination of azacitidine with Venetoclax showed an increased remission rate without improved survival.

Since AML is a highly heterogeneous disease, it is not clear which genetic type of adult AML patients would benefit from Venetoclax combined with intensive chemotherapy.

Therefore, this study intends to conduct a phase II clinical trial to investigate the efficacy of intensive chemotherapy combined with Venetoclax in adult AML patients, and reveal the efficacy of Venetoclax added to chemotherapy regimens for AML with different cytogenetic and molecular subgroups.

DETAILED DESCRIPTION:
Patients will receive 1 course of intensive chemotherapy combined with venetoclax for induction and those who achieved complete remission will receive 3 courses of intermediate-dose cytarabine combined with Venetoclax for consolidation. After consolidation therapy, Venetoclax in combination with azacitidine will be applied for 6 courses as maintenance treatment. Allogeneic hematopoietic stem cell transplantation is recommended for high-risk groups and intermediate-risk with positive measurable residual disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet AML according to WHO (2022) or AML and MDS/AML defined by ICC standards.
2. Age ≥14 years old, ≤ 60 years old, male or female.
3. The physical status assessment (ECOG-PS) of the Eastern Oncology Collaboration group was 0-2 points.
4. Fulfill the requirements of the following laboratory tests (performed within 7 days prior to treatment) :

   1. Total bilirubin ≤ 1.5 times the upper limit of normal value (same age);
   2. AST and ALT≤ 2.5 times the upper limit of normal value (same age);
   3. Blood creatinine < 2 times the upper limit of normal (same age);
   4. Myocardial enzymes < 2 times the upper limit of normal (same age);
   5. Left ventricular ejection fraction >50% by measure of echocardiogram (ECHO). Informed consent must be signed before the commencement of all specific study procedures, and signed by the patient himself or his immediate family. Considering the patient's condition, if the patient's signature is not conducive to the treatment of the condition, the informed consent shall be signed by the legal guardian or the patient's immediate family.

Exclusion Criteria:

Subjects who meet any of the following criteria are excluded from the study:

1. Acute promyelocytic leukemia with PML-RARA fusion gene
2. Acute myeloid leukemia with BCR-ABL fusion gene
3. Treated patients (but can receive hydroxyurea or cytarabine to the lower tumor burden).
4. Concurrent malignant tumors of other organs (those requiring treatment).
5. Active heart disease, defined as one or more of the following:

   1. A history of uncontrolled or symptomatic angina;
   2. Myocardial infarction less than 6 months after enrollment;
   3. Have a history of arrhythmia requiring drug treatment or severe clinical symptoms;
   4. Uncontrolled or symptomatic congestive heart failure (> NYHA level 2);
6. Serious infectious diseases (uncured tuberculosis, pulmonary aspergillosis).
7. Those who were not considered suitable for inclusion by the researchers.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1200 (Estimated)
Dates: Start 2024-09-29 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | up to 2 years after the date of the last enrolled participants
  All patients definitions for the trial; From the date of enrollment to the time of treatment failure after two courses of induction therapy, recurrence after CRc, date of all-cause death, or the date of last survival follow-up.

SECONDARY OUTCOMES:
Complete remission (CR)/CR with partial hematologic recovery (CRh)/CR with incomplete hematologic recovery (CRi) with negative MRD detected by flow cytometry | up to 1 years after the date of the last enrolled participants
  The ratio of CR/CRh/CRi with negative MRD detected by flow cytometry after induction, consolidation, and maintenance therapy.
CR/CRh/CRi with negative MRD detected by PCR | up to 1 years after the date of the last enrolled participants
  The ratio of CR/CRh/CRi with negative MRD detected by PCR after induction, consolidation, and maintenance therapy.
overall survival (OS) | up to 2 years after the date of the last enrolled participants
  Used to evaluate all patients who enter clinical trials. From the date of entry into the trial until the date of patient death (including any cause) or last survival follow-up.
30-day mortality | within 30 days of the date of the last enrolled participants
  Percentage of patients who died within 30 days from enrollment.
60-day mortality | within 60 days of the date of the last enrolled participants
  Percentage of patients who died within 60 days from enrollment.
Complete remission (CR)/CR with partial hematologic recovery (CRh)/CR with incomplete hematologic recovery (CRi) rate | up to 3 months after the date of the last enrolled participants
  The ratio of patients achieved CR/CRh/CRi after two courses of induction therapy.
Relapse-free survival (RFS) | up to 2 years after the date of the last enrolled participants
  Defined only for patients achieving CRc; measured from the date of achievement of remission until the date of hematologic relapse or death from any cause; patients not known to have relapsed or died at last follow-up are censored on the date they were last known to be alive

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wei, MD, Principal Investigator — Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- Blood Diseases Hospital, Tianjin, Tianjin Municipality, China